CLINICAL TRIAL: NCT00000497
Title: Dietary Intervention Study for Hypertension (DISH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 16; U01HL037854 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2000-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases | interventions — Diet, Sodium-Restricted; Diet, Reducing

INTERVENTIONS:
Behavioral: diet, sodium-restricted
Behavioral: diet, reducing

SUMMARY:
The primary objective of this multicenter cooperative clinical trial was to determine if dietary modification would enable drug controlled hypertensive patients to remain at 'goal blood pressures' after antihypertensive medication was withdrawn. The proposal made use of the HDFP hypertensive population who had five years of treatment for their hypertension. Additionally, the group of investigators proposed to determine if dietary treatment would permit patients not previously adequately controlled under the HDFP program to achieve normalization of blood pressure with a combination of dietary modification and drug treatment. The study also proposed to search for predictors (i.e., levels of hormonal agents such as plasma renin activity) of responsiveness to dietary manipulation among the hypertensive population as well as to identify psychological attributes that might be of importance in managing these patients.

DETAILED DESCRIPTION:
BACKGROUND:

The background against which the proposal was made had been developed from the combined information of the Veterans Administration Cooperative Study and the Hypertension Detection and Follow-up Study. Data from both these studies clearly established the importance of reducing sodium content by means of diuretic administration as a mainstay of the treatment of elevated blood pressure. The risks of the lifetime of treatment were undefined, but the cost of indefinite treatment of high blood pressure was sufficiently high to stimulate careful examination of alternative modes of management of such patients. The demonstrations by Parijs and others that moderate reduction in sodium intake led to improved management of hypertension and data suggesting that increased potassium intake may enhance this blood pressure lowering effect associated with sodium restriction was cited by the investigators as a basis for the trial. Any additional data regarding modest sodium restriction and potassium ingestion would have impact on utilizing such therapy in preventing hypertension and as adjunctive therapy.

DESIGN NARRATIVE:

The study was intended to take advantage of the availability of patients at the three centers at the completion of the Hypertension Detection and Follow-up Program Study. These patients were enrolled as 'stepped-care' participants and had been treated with antihypertensive drugs for at least five years. The main objective of the study was to determine the contribution of dietary modification to maintenance of normal blood pressure after withdrawal of medication. Two types of diet change were followed: 1) reduction of sodium intake coupled with increased potassium intake; and 2) reduction of weight in the subgroups of patients that were obese.

ELIGIBILITY:
Men and women with hypertension. Diastolic blood pressure equal to or above 95 mm Hg and 90 mm Hg, respectively for home and clinic readings.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1980-01; Study Completion 1994-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Langford — University of Mississippi Medical Center

REFERENCES:
- [Background] Wassertheil-Smoller S, Langford HG, Blaufox, MD, et al: Rate of Hypertension Return After Withdrawal of Prolonged Antihypertensive Therapy. Clin Sci, 63: 423S-525S (Supp 8), 1982.
- [Background] Wassertheil-Smoller, Langford HG, Blaufox MD, Oberman A, Hawkins M. Diuretics and salt restriction in blood pressure control. Curr Concepts Nutr. 1983;12:175-89. No abstract available. PMID 6342972
- [Background] Langford HG, Blaufox, MD, Oberman A, et al: Effect of Weight Loss on the Return of Hypertension After Withdrawal of Prolonged Antihypertensive Therapy. Nutritional Prevention of Cardiovascular Disease, 301-315, 1984.
- [Background] Wing RR, Caggiula AW, Nowalk MP, Koeske R, Lee S, Langford H. Dietary approaches to the reduction of blood pressure: the independence of weight and sodium/potassium interventions. Prev Med. 1984 May;13(3):233-44. doi: 10.1016/0091-7435(84)90081-1. PMID 6494106
- [Background] Langford HG, Blaufox MD, Oberman A, Hawkins CM, Curb JD, Cutter GR, Wassertheil-Smoller S, Pressel S, Babcock C, Abernethy JD, et al. Dietary therapy slows the return of hypertension after stopping prolonged medication. JAMA. 1985 Feb 1;253(5):657-64. PMID 3881608
- [Background] Langford HG, Schlundt D, Levine K. Sodium restriction in hypertension. Compr Ther. 1984 Sep;10(9):6-11. PMID 6488753